CLINICAL TRIAL: NCT02028273
Title: Hippocampal Neurogenesis in Human Subjects (Pilot Study)
Brief Title: Hippocampal Neurogenesis in Human Subjects
Acronym: NG
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 032012-021
Record Dates: First submitted 2013-01-03; First posted 2014-01-07 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Hippocampal Neurogenesis in Cocaine Addiction
Keywords: Neurogenesis; Addiction; Cocaine; MRI; MRS
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Healthy control group. No history of substance abuse or dependence.
- Actively using patients: Participants actively using cocaine.
- Abstinent Patients: Participants who have been abstinent from cocaine use for 3-6 months.

SUMMARY:
This study is being done to measure the number of brain cells that grow in the brain throughout our lives while determining an effective way to complete this with an MRI (Magnetic Resonance Imaging) scanner. The number of these brain cells may be affected by cocaine use. Researchers are trying to understand the long-term effects of cocaine use on the brain.

DETAILED DESCRIPTION:
New neurons are generated through the process of neurogenesis. Although most active during pre-natal development, neurogenesis persists throughout the human lifespan. In adulthood, neurogenesis occurs predominantly in the subgranular zone of the hippocampal dentate gyrus. A highly novel methodology using Magnetic Resonance Spectroscopy (MRS) has recently been developed to measure the formation of hippocampal newborn stem cells in the human brain. We propose to assess Neural Progenitor Cells (NPCs) in the neuropsychiatric disorder cocaine dependence, a chronic disease process associated with pathology of the hippocampus and impaired neurogenesis. In addition, we will assess other measures associated with neurogenesis, including hippocampal (dentate gyrus) cerebral blood volume (CBV) using Vascular-Space-Occupancy (VASO) Magnetic Resonance Imaging. We predict that newborn hippocampal cells [or neuronal progenitor cells (NPCs] will be attenuated in recently using cocaine-addicted participants relative to abstinent and control participants, and that these changes will be paralleled by changes in CBV. In this pilot study, we will assess for these changes in cocaine-addicted subjects who are actively using cocaine and those who are recently abstinent (three to six months) as well as age-, race-, and gender-similar control participants.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine-dependence (patient population) or no cocaine-dependence (control population)

Exclusion Criteria:

* Other medical or psychiatric disorders that may effect neural functioning
* Medications that may effect neural functioning

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from residential sober living and outpatient facilities. Patients will also be recruited through flyers placed locally. Healthy controls will be recruited from the Greater Dallas community.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Assess Neural Progenitor Cells | within 3 weeks of screening physical
  A 1 hour Magnetic Resonance Spectroscopy to determine the presence of newborn hippocampal neurons in using and abstinent cocaine addicts

SECONDARY OUTCOMES:
Hippocampal cerebral blood volume | within 3 weeks of screening physical
  Measure cerebral blood flow during an hour long Vascular-Space-Occupancy (VASO) Magnetic Resonance Imaging to assess production of hippocampal cells

CONTACTS AND LOCATIONS:
Overall Officials: Bryon Adinoff, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Division on Addictions, Dallas, Texas, United States